CLINICAL TRIAL: NCT01206387
Title: A Double-Blind, Vehicle-Controlled, Randomized, Parallel Design, Multiple-Site Clinical Study to Evaluate the Efficacy and Safety of Desoximetasone 0.25% Topical Spray in Patients With Moderate to Severe Plaque Psoriasis
Brief Title: Effects of Desoximetasone Spray 0.25% on Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DSXS-0808
Record Dates: First submitted 2010-09-20; First posted 2010-09-21 (Estimated); Results first posted 2014-08-07 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-05

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Desoximetasone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- active product (Experimental): Desoximetasone Spray 0.25%
  Interventions: Drug: Desoximetasone Spray 0.25%
- placebo comparator (Placebo Comparator): vehicle
  Interventions: Drug: placebo comparator

INTERVENTIONS:
Drug: Desoximetasone Spray 0.25% — Desoximetasone topical spray 0.25% administered to affected area twice a day for 28 days
  Other Names: Desoximetasone
  Arms: active product
Drug: placebo comparator — Placebo administered to affected area twice a day for 28 days
  Other Names: vehicle
  Arms: placebo comparator

SUMMARY:
efficacy study in patients with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
A Double-Blind, Vehicle-Controlled, Randomized, Parallel Design, Multiple-Site Clinical Study to Evaluate the Efficacy and Safety of Desoximetasone 0.25% Topical Spray in Patients with Moderate to Severe Plaque Psoriasis

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating female 18 years of age or older.
* Have a definite clinical diagnosis of stable plaque psoriasis involving ≥ 10% of the body surface area (BSA).
* Have a combined total lesion severity score (TLSS) of ≥ 7 for the Target Lesion.
* Have a plaque elevation score ≥ 3 of (moderate) for the Target Lesion.
* The Target Lesion must have an area of at least 5 cm².
* Have a Physicians Global Assessment (PGA) score of 3 (moderate) or 4 (severe) at baseline for the overall disease severity.

Exclusion Criteria:

* Patient has current diagnosis of other types of psoriasis other than stable plaque psoriasis (i.e. acute, guttate, erythrodermic, exfoliative or pustular psoriasis) or has psoriasis of any kind of the face or scalp that will require active treatment during the study. Nonprescription antipsoriatic shampoos will be allowed during the study when applied solely to the scalp.
* Patient has a history of psoriasis that has been unresponsive to topical corticosteroid therapy.
* In the Investigator's opinion, the patient has other dermatological conditions, such as atopic or contact dermatitis, that may interfere with the clinical assessments of the signs and symptoms of psoriasis.
* Patient has a history of allergy or sensitivity to corticosteroids or history of any drug hypersensitivity or intolerance which, in the opinion of the Investigator, would compromise the safety of the patient or the results of the study.
* Patient has been treated within 12 weeks (or five half lives, whichever is less) prior to the first dose of study drug with any biological therapies for psoriasis.
* Patient has received any systemic steroids within 4 weeks of the first dose of the study drug. The use of inhaled or intranasal corticosteroids is acceptable as long as usage has been stable for at least 2 weeks prior to the first dose of study drug and will be continued during the study.
* Patients who have used any topical antipsoriatic agents of any kind or any topical corticosteroids for any reason within 2 weeks prior to first use of study drug. Nonprescription antipsoriatic shampoos used only on the scalp will be allowed during the study.
* Receipt of any drug as part of a research study within 30 days prior to first dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-08; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novum Pharmaceutical Research Services, Study Chair — http://www.novumprs.com/contact

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saleem MD, Negus D, Feldman SR. Topical 0.25% desoximetasone spray efficacy for moderate to severe plaque psoriasis: a randomized clinical trial. J Dermatolog Treat. 2018 Feb;29(1):32-35. doi: 10.1080/09546634.2017.1331027. Epub 2017 May 30. PMID 28504031

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: placebo comparator: Placebo administered to affected area twice a day for 28 days
Period: Overall Study
Arm/Group | Desoximetasone Spray 0.25% | Placebo
Started | 60 | 60
Completed | 59 | 60
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Desoximetasone Spray 0.25% | Placebo | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.67 (13.86) | 52.55 (15.56) | 51.61 (14.71)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 14 | 28
  Between 18 and 65 years | 36 | 29 | 65
  >=65 years | 10 | 17 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 42 | 43 | 85
Region of Enrollment [Number; unit: participants]
  United States | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Clinical Success
Description: A patient is considered a Clinical Success if the Physician's Global Assessment (PGA) is 0 (clear) or 1 (almost clear).
Time Frame: 28 days
Population: Primary Efficacy Analysis at Day 28 Clinical Success (ITT)
Measure: Number; unit: participants
Arm/Group | Desoximetasone Spray 0.25% | Placebo
Number analyzed (Participants) | 59 | 60
participants | 18 | 3
Statistical Analysis 1: Comparison: Desoximetasone Spray 0.25% vs Placebo; Test type: Superiority or Other; p = 0.0003, t-test, 2 sided

2. Primary Outcome: Treatment Success
Description: A patient is considered a Treatment Success for the Target Lesions if the target lesion has a score of 0 or 1 on the Target Lesion Severity Score (TLSS)for each of each of the three signs and symptoms (erythema, scaling and plaque elevation).
Time Frame: 28 days
Measure: Number; unit: participants
Arm/Group | Desoximetasone Spray 0.25% | Placebo
Number analyzed (Participants) | 59 | 60
participants | 23 | 4
Statistical Analysis 1: Comparison: Desoximetasone Spray 0.25% vs Placebo; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

3. Secondary Outcome: Mean Change From Baseline in Physician Global Assessment (PGA) Score at Day 28 Using ITT.
Description: In the Physician Global Assessment of psoriasis is a score based on physician assessment of overall disease severity for all lesions assessed at baseline and at Day 28. The PGA score range: from 0 (Clear=No Psoriatic lesions, i.e. no plaque formation; no erythema, no induration, no scaling) to 5 (Very Severe=Coarse scaling with pronounced cracking and fissures. Erythema is dark red with induration. Plaques are markedly elevated with sharp and hard edges).
  The first evaluation was for the change from baseline in PGA, using a two-sided, α = 0.05 level of significance. If superiority of the test product over its vehicle was demonstrated (p<0.05), then PGA change from baseline values was examined.
Time Frame: Baseline and day 28
Population: All participants enrolled in this study were included in this intent-to-treat (ITT) analysis. Results are presented as observed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Desoximetasone Spray 0.25% | Placebo
Number analyzed (Participants) | 59 | 60
units on a scale | 1.14 (0.9) | 0.50 (0.68)
Statistical Analysis 1: Comparison: Desoximetasone Spray 0.25% vs Placebo; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

4. Secondary Outcome: Mean Change From Baseline in Total Lesion Severity Scale (TLSS) (ITT)
Description: Mean Change from Baseline in Lesion Severity Scale-TLSS (ITT)
  TLSS of psoriasis is a combined score based on physician assessment of disease severity for the Target Lesion assessed at baseline and at Day 28. The TLSS combined score included summary of individually scored induration (as 0=Clear or 1=Almost Clear, or 2=Mild, or 3=Moderate, or 4=Severe, or 5=Very Severe), erythema (as 0=Clear or 1=Almost Clear, or 2=Mild, or 3=Moderate, or 4=Severe, or 5=Very Severe), and scaling (as 0=Clear or 1=Almost Clear, or 2=Mild, or 3=Moderate, or 4=Severe, or 5=Very Severe). To be eligible for inclusion in the study, the combined score of all three signs for the Target Lesion must total at least 7 and the patient must have at least a score of 3=Moderate for plaque elevation
  The first evaluation was for the change from baseline in TLSS, using a two-sided, α = 0.05 level of significance.
Time Frame: Baseline and day 28
Population: Base on intention to treat. All participant with mean change from baseline in TLSS at Day 28
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Desoximetasone Spray 0.25% | Placebo
Number analyzed (Participants) | 59 | 60
units on a scale | 4.73 (3.08) | 1.93 (1.96)
Statistical Analysis 1: Comparison: Desoximetasone Spray 0.25% vs Placebo; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

5. Secondary Outcome: Mean Change From Baseline in Percent Body Surface Area (%BSA) Affected at Day 28
Description: Mean Change from Baseline in percent body surface area (%BSA) affected by Psoriasis
  The Body Surface Area (BSA) is a numerical score used to measure the physician's assessment of the percentage of the participant's total BSA involved with psoriasis.
  BSA = SQRT ((height (cm) X weight (kg))/3600) BSA is in m2, W is weight in kg, and H is height in cm. Total body Surface Area (BSA) in meters squared
  For the %Body Surface Area Affected the "Rule of Nine" was be used.
  Change From Baseline in Percent Body Surface Area i.e., difference of base percent values [Percent Body Surface Area at 28 days - Percent Body Surface Area at Baseline].
Time Frame: Baseline and day 28
Population: Base on intention to treat. All participant with Mean Change from Baseline in %BSA affected at Day 28
Measure: Mean (Standard Deviation); unit: percentage of body surface area affected
Arm/Group | Desoximetasone Spray 0.25% | Placebo
Number analyzed (Participants) | 59 | 60
percentage of body surface area affected | 2.24 (3.79) | 0.37 (2.05)
Statistical Analysis 1: Comparison: Desoximetasone Spray 0.25% vs Placebo; Test type: Superiority or Other; p = 0.0011, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 3 months
Description: Daily questionnaire
Arm/Group | Desoximetasone Spray 0.25% | Placebo
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 17/60 | 21/60
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Desoximetasone Spray 0.25% (N=60) | Placebo (N=60)
Application Site Dryness (Skin and subcutaneous tissue disorders) | 4 (7) | 5 (6)
Application Site Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Application Site Irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Application Site Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 6 (6)
Arthralgia (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 3 (5) | 1 (3)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Sinus Headache (Nervous system disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No